CLINICAL TRIAL: NCT00352820
Title: The Experience of Informal Caregivers of Patients With Brain Tumors
Brief Title: Experience of Brain Tumor Caregivers
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0019
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Brain Cancer; Glioma
Keywords: Caregiver; Brain cancer; Glioma; Questionnaire; Survey; Interview
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interview + Questionnaire
  Interventions: Behavioral: Interview; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Interview — Recorded face-to-face session.
Behavioral: Questionnaire — Written survey lasting approximately 30 minutes.
  Other Names: Survey

SUMMARY:
The objective of this study is to explore the experience of informal caregivers of patients with a primary brain tumor, identifying elements and themes of the caregiving experience specific to this population of caregivers. The aim is to describe the experience of being an informal caregiver for a patient with a primary brain tumor.

DETAILED DESCRIPTION:
Caregiver Consent:

If you agree to take part in this study, you will be asked to have 1 interview. This will be a face-to-face interview that will take place at M. D. Anderson while you are there for the patient's physician appointment.

During this interview, you will be asked to describe what it has been like for you to help care for a person with a primary brain tumor in the past, what it is like to care for a person with a primary brain tumor now, and what you think it might be like in the future. You will be interviewed alone, and your interview will be tape recorded and then written on paper. The information that is gathered (the tape and the written information) will be kept strictly confidential. The tapes and any paperwork will be kept in a locked box during and after this study. The written information will be kept in password-protected computer files. The researcher is the only person who will have access to the tapes. You will also be asked to answer a questionnaire on paper. This questionnaire will ask specific personal information, such as your age, occupation, and relationship to the patient. This questionnaire will take about 5 minutes to complete. The entire interview will take about 30 minutes to complete.

Your participation in this study will be over after you complete the interview and the questionnaire.

This is an investigational study. Up to 20 caregivers will take part in this study. All will be enrolled at M. D. Anderson.

Patient Consent:

If you agree to take part in this study, you will be asked to choose a family member or a friend who is your main caregiver and who may be willing to take part in 1 interview for this study. Your consent in this study, will give researchers permission to contact your caregiver. If your caregiver chooses to participate, the interview will be face-to-face, and it will take place at M. D. Anderson while you are there for your physician appointment. During this interview, the caregiver will be asked to describe what it has been like for them to help care for you. The researcher will get informed consent from your caregiver and will go into further detail about this study.

He or she will be interviewed alone, and the information gathered during the interview will be kept strictly confidential. Your caregiver will be asked to complete a questionnaire for specific personal information, such as his or her age, occupation, and relationship to you. The entire interview will take about 30 minutes to complete.

You will be asked to allow your sociodemographic data (such as your gender, marital status, etc.) and medical data (such as your diagnosis, therapies received, etc.) to be collected from your medical record. This information will be used to help researchers learn about the unique backgrounds of the patients participating in this study. Your information that is gathered will be kept strictly confidential, and it will be kept in a locked box during and after this study.

Your participation in this study will be over after your sociodemographic and medical data have been collected from your medical record.

This is an investigational study. Up to 20 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Ability to speak and read English
3. Diagnosis of a primary brain glioma, World Health Organization Grade II-IV (PATIENT ONLY)
4. At least 3 months since time of diagnosis (PATIENT ONLY)
5. Identification as the primary informal caregiver by a patient with a primary brain glioma (CAREGIVER ONLY)
6. Consent to participate

Exclusion Criteria:

1. Inability to understand the intent of the study
2. Medical condition that would preclude participation in an interview lasting 30 minutes (CAREGIVER ONLY)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary informal caregiver of individual with a primary brain glioma.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Descriptive exploratory analysis to identify themes and describe experience of caring for a person with a primary brain tumor | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Loretta A. Williams, DSN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org